CLINICAL TRIAL: NCT01808781
Title: The Effect of Home-Based High-Velocity Training on Muscle Strength and Power, Functional Performance, and Physical Activity Behavior in Individuals With Total Knee Arthroplasty.
Brief Title: The Effect of Home-based Velocity Training in Individuals With Total Knee Replacement
Acronym: TKR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Texas Physical Therapy Association (Other)
Responsible Party: Principal Investigator, Emerenciana Hines, PhD Student, Texas Woman's University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 17263
Record Dates: First submitted 2013-03-06; First posted 2013-03-11 (Estimated); Last update posted 2017-10-12 (Actual); Status verified 2017-10

CONDITIONS: Total Knee Arthroplasty
Keywords: Power; muscle strength; total knee replacement; physical activity behavior
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Home exercise program plus walking program during 8-week period
  Interventions: Other: Exercises plus walking program
- Comparison group (Active Comparator): Walking only program throughout the 8-week period.
  Interventions: Other: Walking only program

INTERVENTIONS:
Other: Exercises plus walking program — Exercise group Consist of functional exercises such as mini-squats, sit to stand, and exercises with use of thera-bands. For each exercise, participants will be taught to perform the concentric phase forcefully and as fast as they can and return to the initial position slowly and with control. Participants will be asked to perform the exercises 3 times per week as a home exercise program daily throughout the 8-week intervention period. Additionally, they will be asked to wear a pedometer daily throughout the 8-week intervention to monitor steps. A step goal will be provided to gradually increase daily to become "somewhat active" or "active" by the end of the 8-week intervention.
  Arms: Intervention group
Other: Walking only program — Participants will be asked to wear a pedometer and instructions for use just as the exercise group. They will also will given a step goal just as the participants in the exercise group and will similarly be asked to record number of steps form their pedometer in a daily log along with the minutes of moderate and vigorous physical activity throughout the 8-week intervention period.
  Arms: Comparison group

SUMMARY:
The purpose of this study will be to find out the effect of two different interventions on muscle strength, ability to produce muscle force quickly (power), daily function, and number of steps and physical activity an individual with total knee replacement do daily.

The research hypotheses for this study will be as follows:

* For individuals who are at least 6 months post-total knee replacement, home-based high-velocity training exercises will result in significantly greater improvements in muscle strength and power compared to those who receive a walking program only.
* For individuals who are at least 6 months post-total knee replacement, home based high-velocity training exercises will result in significantly greater improvements of daily function(eg. sit to stand, climb a set of stairs)than those who receive a walking program only.
* For individuals who are at least 6 months post-total knee replacement, home based high-velocity training exercises will result in significantly greater improvements in physical activity behavior (eg. number of steps per day)compared to those who receive a walking program only.

ELIGIBILITY:
Inclusion Criteria:

* Men and women who are at least 40 years of age will qualify if they had a primary unilateral total knee replacement (TKR) 6 to 18 months.

Exclusion Criteria:

* other lower extremity prosthetic implants other than the current TKR
* revision TKR or plan for revision
* diagnosis of severe osteoarthritis in the uninvolved knee or either hip joints
* recent low extremity injury or significant pain that increases during weight bearing or other functional performance
* diagnosis of neurologic deficits
* decreased cognitive status that might affect the ability to follow instructions
* significant cardiovascular and/or pulmonary disease that limits function

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
Muscle Power | Baseline and 8 weeks
  Change in quadriceps muscle power (force versus velocity)

SECONDARY OUTCOMES:
muscle strength | Baseline and 8 weeks
  Change in quadriceps muscle strength.

OTHER OUTCOMES:
Functional Performance | Baseline and 8 weeks
  Change the ability to perform the stair climb test faster and walking a further distance during the 6 minute walking test.
Physical activity behavior | Baseline and 8 weeks
  increase the number of steps per day and the minutes of moderate and/or vigorous physical activities.

CONTACTS AND LOCATIONS:
Overall Officials: Emerenciana S Hines, PhD, Principal Investigator — Texas Woman's University
Locations (1):
- Texas Woman's University, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We are planing to publish the results and sharing all the data with a journal interested in this study.

REFERENCES:
- [Derived] Trudelle-Jackson E, Hines E, Medley A, Thompson M. Exploration of Habitual Walking Behavior and Home-Based Muscle Power Training in Individuals With Total Knee Arthroplasty. J Phys Act Health. 2020 Mar 1;17(3):331-338. doi: 10.1123/jpah.2019-0233. PMID 32023537